CLINICAL TRIAL: NCT01681771
Title: Internet Cognitive Behavioural Therapy to Patients With Heart Failure and Depression A Randomised Controlled Study of Short and Long Term Effects on Depressive Symptoms
Brief Title: Internet Cognitive Behavioural Therapy to Patients With Heart Failure and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Peter Johansson, Nurse, Assoc. Prof, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORSS-221791
Record Dates: First submitted 2012-08-30; First posted 2012-09-10 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure; Depressive Symptoms
MeSH Terms: conditions — Heart Failure; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cogntive behaviour therapy (Experimental): Internet based Cognitive behaviour therapy during 9 weeks
  Interventions: Behavioral: Cognitive behaviour therapy
- Discussion group (Active Comparator): Internet moderated discussion group during 9 weeks
  Interventions: Behavioral: Cognitive behaviour therapy; Behavioral: Discussion group

INTERVENTIONS:
Behavioral: Cognitive behaviour therapy — Internet based, weekly home task and weekly feedback provided by health care professional.
Behavioral: Discussion group — Internet moderated discussion group. Patients will be provided weekly question which will be used by the participant to start discuss with each others.
  Arms: Discussion group

SUMMARY:
The purpose of this study is to evaluate the short (9 weeks) and long (6 and 12 months) term effects of an 9 weeks intervention of internet-based cognitive behavioural therapy on depressive symptoms, worrying/anxiety, sleep, self-care knowledge and quality of life in patients with chronic heart failure and depression.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* have time to participate in the study,
* treatment for HF according to the European Society of Cardiology guidelines2
* stable HF (NYHA class I-III) and not being hospitalized for HF the latest month
* signs of suffering of depressive symptoms (Patient Health Questionnaire-9 >9 points

Exclusion Criteria:

* severe HF (NYHA IV) or another severe chronic life threatening disease.
* severe depression assessed to need hospital care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Johansson, Assoc. Prof, Principal Investigator — Department of Cardiology, University Hospital of Linköping and Department of Cardiovascular Medicine, Faculty of Health Sciences. University Hospital of Linköping
Locations (1):
- Deparment of Cardiology, University Hospital of Linköping, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lundgren JG, Dahlstrom O, Andersson G, Jaarsma T, Karner Kohler A, Johansson P. The Effect of Guided Web-Based Cognitive Behavioral Therapy on Patients With Depressive Symptoms and Heart Failure: A Pilot Randomized Controlled Trial. J Med Internet Res. 2016 Aug 3;18(8):e194. doi: 10.2196/jmir.5556. PMID 27489077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recrutiment from medical clinics
Pre-assignment Details: No pre-assignment details to report
Period: Overall Study
Arm/Group | Cogntive Behaviour Therapy | Discussion Group
Started | 25 | 25
Completed | 21 | 23
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cogntive Behaviour Therapy | Discussion Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (13.9) | 62.3 (11.7) | 62.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms
Description: Depressive Symptoms measured with Patient Health Questionnaire-9 (PHQ-9). The number of patients per study arm is planned to be n=60. According to an earlier metaanalysis, the effect size of internet CBT intervention can be expected to be at least at the level of 0.5. The score on the PHQ-9 ranges from 0-27. A score between 5-10 indicate a mild depression whereas a score >10 indicate at least moderate depression.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cogntive Behaviour Therapy | Discussion Group
Number analyzed (Participants) | 25 | 25
units on a scale | 8.6 (4.6) | 9.8 (4.3)
Statistical Analysis 1: Comparison: Cogntive Behaviour Therapy vs Discussion Group; Test type: Superiority; p = 0.21, ANCOVA; ANCOVA analysis comparing PHQ-9 mean values at 9 weeks follow-up between the I-CBT and discussion group and adjusting for PHQ-9 values baseline

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: Weekly measurement of depression to asses if participants depression not deteroriated and became severe requiring contact with a health care providor
Arm/Group | Cognitive Behavoural Therapy | Discussion Group
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No